CLINICAL TRIAL: NCT05349435
Title: A Phase 1, Randomised, Open-Label, Crossover Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Ascending Doses of PBI-4050 Compared to Sodium Phenylbutyrate in Healthy Subjects
Brief Title: A Healthy Volunteer Study to Compare Fezagepras (PBI-4050) With Sodium Phenylbutyrate
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor has decided to discontinue development of fezegepras based on initial pharmacokinetic results
Sponsor: Liminal BioSciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PBI-4050-CT-9-21
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Hyperammonemia
MeSH Terms: conditions — Hyperammonemia | interventions — setogepram; 4-phenylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 Dose Level 1 (Experimental): Drug: Fezagepras and sodium PBA
  Interventions: Drug: Fezagepras; Drug: Sodium phenylbutyrate
- Cohort 2 Dose Level 2 (Experimental): Drug: Fezagepras and sodium PBA
  Interventions: Drug: Fezagepras; Drug: Sodium phenylbutyrate

INTERVENTIONS:
Drug: Fezagepras — Investigational drug
  Other Names: PBI-4050
Drug: Sodium phenylbutyrate — Investigational drug

SUMMARY:
The purpose of this study is to compare the safety, tolerability and pharmacokinetic profile of fezagepras (PBI-4050) to that of sodium phenylbutyrate (PBA) when both products are given as single ascending doses to healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female (of non childbearing potential only*), 18 to 65 years of age, inclusive, at the screening visit.

   * Females of childbearing potential are defined as fertile, following menarche and until becoming post menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
   * Females of non-childbearing potential are defined as females who have undergone a sterilization procedure at least 6 months prior to the first dosing or females who are postmenopausal.
2. Male subjects must follow protocol specified contraception guidance
3. Continuous non smoker who has not used nicotine and tobacco containing products for at least 3 months prior to the first dosing based on subject self-reporting.
4. Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2 and body weight of ≥ 50 kg for males and ≥ 45.0 kg for females, at the screening visit.
5. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs and ECGs, as deemed by the PI or designee, including the following:

   * Seated blood pressure is ≥ 90/40 mmHg and ≤ 140/90 mmHg at the screening visit.
   * Seated heart rate is ≥ 40 bpm and ≤ 99 bpm at the screening visit.
   * QTcF interval is ≤ 460 msec (males) and ≤ 470 msec (females) and has ECG findings considered normal or not clinically significant by the PI or designee at the screening visit.
   * Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min at the screening visit.
   * Hemoglobin ≥ 128 g/L (males) or ≥ 115 g/L (females) and hematocrit ≥ 0.36 L/L (males) or ≥ 0.32 L/L (females) at screening.
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ upper limit of normal (ULN), total bilirubin ≤ 2 ULN or creatinine is ≤ ULN.
6. Able to swallow multiple tablets.
7. Understands the study procedures in the informed consent form (ICF), able to provide written consent and be willing and able to comply with the protocol to completion of the study (including follow-up visit).

Exclusion Criteria:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease, including but not limited to neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. History of any illness that might confound the results of the study or pose an additional risk to the subject by their participation in the study.
4. History of significant drug abuse within 18 months prior to screening or use of soft drugs (such as marijuana) within 6 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine, crack, opioid derivatives including heroin, and amphetamine derivatives) within 18 months prior to screening.
5. Drink alcohol in excess of 21 units per week for males or 14 glasses/units per week for females, with one unit = 150 mL of wine or 360 mL of beer or 45 mL of 45% alcohol.
6. History or presence of hypersensitivity or idiosyncratic reaction to the study drug(s) or related compounds.
7. History or presence of:

   * Clinically significant allergic reactions (e.g., anaphylactic reaction and angioedema) to any drug at the discretion of the PI or designee.
   * Clinically significant illness or surgery within 4 weeks prior to dosing at the discretion of the PI or designee. Subjects vomiting within 24 hours pre-dose will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the PI or designee.
8. Female subjects of childbearing potential.
9. Female subject with a positive pregnancy test at the screening visit or at check in or who are lactating.
10. Positive urine drug or alcohol results at the screening visit or check in.
11. Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at the screening visit.
12. Unable to refrain from or anticipates the use of:

    * Over-the-counter products and natural health products (including herbal remedies, homeopathic medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to dosing
    * Any drugs, including prescription and non prescription medications beginning 14 days prior to the first dosing.
    * Any drugs known to be significant inducers of CYP2C9 enzymes and/or P-gp, including St. John's Wort, for 28 days prior to the first dosing
    * Any depot injection or an implant of any drug within 3 months prior to first dosing.
13. Has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 30 days prior to the first dosing.
14. Donation of blood (e.g approximately 500 mL) or plasma within 60 days prior to the first dosing.
15. Donation of bone marrow within the last 6 months prior to the first dosing.
16. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first (if applicable) dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first (if applicable) dosing, or concomitant participation in an investigational study involving no drug or device administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Day -2 to Day 8 (+/- 3 days)
  Number and Severity of Treatment Emergent Adverse Events

SECONDARY OUTCOMES:
AUC | Day 1 and Day 3
  Area under the concentration-time curve
Cmax | Day 1 and Day 3
  Maximum plasma concentration
Tmax | Day 1 and Day 3
  Time to reach maximum plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Sami Omar, Study Director — Liminal BioSciences Ltd.
Locations (1):
- Celerion, Belfast, Northern Ireland, United Kingdom